CLINICAL TRIAL: NCT01785654
Title: Hemodynamic and Biological Evaluations During Reventilation Collapse in ICU
Acronym: REVECOL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0142; DC-2012-1501
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Arterial Line; Consent of Patients; Adult Patients; Tracheal Intubation in ICU
Keywords: Reventilation collapse; Rate of reventilation collapse; Risk factor of reventilation collapse; Hemodynamic profile of reventilation collapse; Biologic approach of reventilation collapse

GROUPS / COHORTS (1):
- reventilation collapse

SUMMARY:
Prospective, observational clinical multicentric study in ICU; during the period surrounding the orotracheal intubation.

DETAILED DESCRIPTION:
Main objective: to describe the characteristics of reventilation collapse: collapse rate, duration and treatment implemented

Secondary objectives:

* identify risk factors of reventilation collapse
* compare mortality, hemodynamic, respiratory, infectious and biological data between collapse group and no reventilation collapse group.

ELIGIBILITY:
Inclusion Criteria:

* Arterial line
* Consent of patients
* Adult patients
* Tracheal intubation in ICU

Exclusion Criteria:

* tracheal intubation for cardiac arrest
* pregnant woman
* major protected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Defined population
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Reventilation collapse | at day 1 (at least thirty minutes despite 500 or 1000ml of fluid resuscitation)

SECONDARY OUTCOMES:
reventilation collapse | in the last 72 hours
Duration of mechanical ventilation | at day 1
mortality | at day 28

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France